CLINICAL TRIAL: NCT02022007
Title: Metabolic and Endocrine Effects of Combination of Metformin and DPP-4 Inhibitor Saxagliptin Compared to Saxagliptin or Metformin XR Monotherapy in Patients With PCOS and Impaired Glucose Regulation: A Single-blinded Randomized Pilot Study
Brief Title: Saxagliptin + Metformin Compared to Saxagliptin or Metformin Monotherapy in PCOS Women With Impaired Glucose Homeostasis
Acronym: BMS-AZPCOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Woman's (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Karen Elkind-Hirsch, Director of Research, Woman's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP13-013; BMS CV181-354 (Other Grant/Funding Number: Bristol Myers Squibb/Astra Zaneca)
Record Dates: First submitted 2013-12-17; First posted 2013-12-27 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Polycystic Ovary Syndrome; Disorder of Glucose Regulation
Keywords: PCOS; IGT; DPP-4 inhibitor
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; saxagliptin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metformin XR (Active Comparator): Metformin 2000 mg daily (QD) for 16 weeks
  Interventions: Drug: Metformin XR
- Saxagliptin (Active Comparator): Saxagliptin 5 mg QD for 16 weeks
  Interventions: Drug: Saxagliptin
- Saxagliptin-Metformin XR (Experimental): Saxagliptin-Metformin XR (combination pill)
  5mg Saxagliptin/2000 mg Metformin XR QD for 16 weeks
  Interventions: Drug: Saxagliptin-Metformin XR

INTERVENTIONS:
Drug: Metformin XR — Start 2 pills (2 pills of 500 mg =1000mg XR) for 3 weeks
  Increase to 4 pills as tolerated (4 pills of 500 mg XR =2000 mg XR) for remainder of study
  Other Names: Glucophage XR; Biguanide-insulin sensitizer
  Arms: Metformin XR
Drug: Saxagliptin — Start 1 pill (5 mg)) for 3 weeks
  Remain at 1 pill (5mg dose) for remainder of study
  Other Names: Onglyza; DPP-4 inhibitor
  Arms: Saxagliptin
Drug: Saxagliptin-Metformin XR — Start 1 pill (2.5 mg/ 1000mg XR) for 3 weeks
  Increase to 2 pills as tolerated (5mg/2000 mg XR) for remainder of study
  Other Names: Kombiglyze XR; Combination DPP-4 inhibitor and Glucophage XR
  Arms: Saxagliptin-Metformin XR

SUMMARY:
The objective of the present proposal is to compare the clinical, endocrine and metabolic effects of therapy with combination saxagliptin and metformin to saxagliptin and metformin monotherapy in women with PCOS and prediabetic hyperglycemia (IFG, IGT or IFG/IGT). Saxagliptin is an oral dipeptidyl peptidase IV (DPP-4) inhibitor whose mechanism of action is to prolong the duration of blood glucagon-like peptide (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP) levels by inhibiting their degradation and thereby augmenting insulin secretion. This study will serve as a pilot investigation to open perspectives for future studies to explore the potential of combining anti-diabetic drugs with different mechanisms of action in in patients with PCOS and impaired glucose regulation (IGR), especially ones for whom standard treatment with metformin is less effective.

DETAILED DESCRIPTION:
A major change in the treatment of polycystic ovary syndrome (PCOS) was initiated by the understanding that many women with this disorder compensate insulin resistance with a period of hypersecretion of insulin by the pancreatic ß-cell. In addition, women with PCOS have significantly higher basal insulin secretory rates, reduced insulin clearance rates, and attenuated secretory responses to meals. The decreased postprandial response in these patients resembles the ß-cell dysfunction of type 2 diabetes (DM2) and may account for the increased incidence of impaired glucose tolerance in this population. Current research has shown that the use of diabetes management practices aimed at reducing insulin resistance and hyperinsulinemia (such as weight reduction and the administration of oral antidiabetic drugs) in women with PCOS can not only improve glucose and lipid metabolism but can also reverse testosterone abnormalities and restore menstrual cycles.

The optimal modality for long-term treatment of PCOS should positively influence androgen synthesis, sex hormone binding globulin (SHBG) production, the lipid profile, insulin sensitivity, and clinical symptoms including hirsutism and irregular menstrual cycles. Improvement of insulin sensitivity may reverse some of the demand on the ß-cell and promote improvement in glucose tolerance. However, while insulin resistance plays a key role in the predisposition to diabetes in PCOS; defects in insulin secretion also appear to contribute to its development. Preferably therapy for women with PCOS should also produce no weight gain, hypoglycemia, or other limiting or unmanageable side effects as well as preserve or enhance ß-cell function.

Presently, in the literature, there are described new, more efficient methods of diabetes prevention in groups with a high risk of this disorder, which involve both, lifestyle modification and pharmacological therapies. Lifestyle intervention was found to reduce the incidence of type 2 diabetes by 58% and metformin by 31% as compared with placebo. The use of rosiglitazone in subjects with prediabetes resulted in a 60% reduction of the diabetes incidence rate. Whether pharmacological therapy should be prescribed for diabetes prevention is an open question given that waiting to add drug therapy until diabetes develops can arrest β-cell decline, albeit at a lower level of β-cell function than when medications are used for prevention. Studies are needed for optimal postpartum and long-term health of women who have had gestational diabetes (GDM). Considerable recent evidence suggests that incretin-based therapies may be useful for the prevention of DM2. Whereas native GLP-1 has a very short half-life, continuous infusion of GLP-1 improves first and second-phase insulin secretion suggesting that early GLP-1 therapy may preserve ß-cell function in subjects with IGT or mild DM2. Incretin mimetics and inhibitors of the protease dipeptidyl peptidase (DPP)-4 use the anti-diabetic properties of the incretin hormone, glucagon-like peptide (GLP)-1 hormone to augment glucose-induced insulin secretion in a highly glucose-dependent manner, thus preventing GLP-1 alone from provoking hypoglycemia. Additional beneficial effects of GLP-1 on endocrine pancreatic islets are that it 1) supports the synthesis of proinsulin to replenish insulin stores in β-cells; 2) reduces the rate of β-cell apoptosis when islets are incubated in a toxic environment (glucotoxicity, lipotoxicity, cytotoxic cytokines); and 3) promotes differentiation of precursor cells with the ability to develop into β-cells and proliferation of β-cell lines, and in whole animals (rodent studies), this leads to an increased β-cell mass within a few days or weeks. Furthermore, GLP-1 can lower glucagon concentrations, i.e., induce α-cells to respond again to the inhibitory action of hyperglycemia, while leaving the counterregulatory glucagon responses undisturbed, as in the case of hypoglycemia. Additional activities of GLP-1 are the deceleration of gastric emptying, which slows the entry of nutrients into the circulation after meals, a reduction in appetite, and earlier induction of satiety, leading to weight reduction with chronic exposure. Inhibition of DPP-4 increases the concentration of GLP-1 and may potentially delay disease progression in prediabetes considering the β-cell function improvement in DM2 and β-cell mass shown to increase in animal models. The objective of the present proposal is to compare the clinical, endocrine and metabolic effects of therapy with combination saxagliptin and metformin to saxagliptin and metformin monotherapy in women with PCOS and prediabetic hyperglycemia (IFG, IGT or IFG/IGT). Since aberrant first-phase insulin secretion and impaired suppression of endogenous glucose production are major contributors to postprandial hyperglycemia and development of DM2, the effects of saxagliptin to target these defects, and normalize glucose excursions are likely to be clinically significant in patients with PCOS and impaired glucose regulation. This study will evaluate the impact of treatment with combination of metformin and saxagliptin (Kombiglyze XR) compared to saxagliptin (Onglyza) or metformin XR (Glucophage XR) monotherapy over a 16-week period on glycemia and insulin action (fasting, 2 hour, and mean stimulated glucose levels, insulin sensitivity and secretion), hyperandrogenism (total T, DHEAS, SHBG and calculated free androgen index [FAI]), cardiometabolic markers (lipid profile, blood pressure), and anthropometric measurements (BMI, waist: hip ratio, absolute weight) in patients with PCOS and prediabetic hyperglycemia

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years to 42 years of age with polycystic ovary syndrome(NIH PCOS criteria) with prediabetic hyperglycemia determined by an 75 gram oral glucose tolerance test (OGTT). Study subjects will be inclusive of PCOS women with impaired fasting glucose (IFG), impaired glucose tolerance (IGT), or both (IFG/IGT).
* Written consent for participation in the study

Exclusion Criteria:

* Presence of significant systemic disease, heart problems including congestive heart failure, history of pancreatitis, or diabetes mellitus (Type 1 or 2)
* Any hepatic diseases in the past (viral hepatitis, toxic hepatic damage, jaundice of unknown etiology), gallstones, abnormal liver function tests or renal impairment (elevated serum creatinine levels or abnormal creatinine clearance)
* Uncontrolled thyroid disease (documented normal TSH), Cushing's syndrome, congenital adrenal hyperplasia or hyperprolactinemia
* Significantly elevated triglyceride levels (fasting triglyceride > 400 mg %)
* Untreated or poorly controlled hypertension (sitting blood pressure > 160/95 mm Hg)
* Use of hormonal medications, drugs known to affect gastrointestinal motility, lipid-lowering (statins, etc.) and/or anti-obesity drugs or medications that interfere with carbohydrate metabolism (such as isotretinoin, hormonal contraceptives, gonadotropin releasing hormone (GnRH) analogues, glucocorticoids, anabolic steroids, C-19 progestins) for at least 8 weeks. Use of anti-androgens that act peripherally to reduce hirsutism such as 5-alpha reductase inhibitors (finasteride, spironolactone, flutamide) for at least 4 weeks
* Prior history of a malignant disease requiring chemotherapy
* Known hypersensitivity or contraindications to use of insulin sensitizers such as metformin or thiazolidinediones
* History of hypersensitivity reaction to saxagliptin or other DPP-4 inhibitors (e.g. anaphylaxis, angioedema, exfoliative skin conditions)
* Current use of metformin, thiazolidinediones, glucagon-like peptide -1 receptor agonists, DPP-4 inhibitors, or weight loss medications (prescription or OTC) Patients must stop use of insulin sensitizers or antidiabetic medicines such as metformin for at least 4 weeks or thiazolidinediones, GLP1 agonists or DPPIV inhibitors for 8 weeks.
* Prior use of medication to treat diabetes except gestational diabetes
* Use of drugs known to exacerbate glucose tolerance
* Eating disorders (anorexia, bulimia) or gastrointestinal disorders
* Suspected pregnancy (documented negative serum pregnancy test), desiring pregnancy during the study treatment interval, breastfeeding, or known pregnancy in last 2 months
* Active or prior history of substance abuse (smoke or tobacco use within past 3 years) or significant intake of alcohol or history of alcoholism
* Patient not willing to use adequate barrier contraception during study period (unless sterilized or have an IUD).
* Debilitating psychiatric disorder such as psychosis or neurological condition that might confound outcome variables
* Inability or refusal to comply with protocol
* Not currently participating or having participated in an experimental drug study in previous three months

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Elkind-Hirsch, Ph.D., Principal Investigator — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elkind-Hirsch KE, Paterson MS, Seidemann EL, Gutowski HC. Short-term therapy with combination dipeptidyl peptidase-4 inhibitor saxagliptin/metformin extended release (XR) is superior to saxagliptin or metformin XR monotherapy in prediabetic women with polycystic ovary syndrome: a single-blind, randomized, pilot study. Fertil Steril. 2017 Jan;107(1):253-260.e1. doi: 10.1016/j.fertnstert.2016.09.023. Epub 2016 Oct 27. PMID 28228317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PCOS women age 18 and 42 years and impaired glucose regulation were enrolled in the study from March 2014 to January 2016. PCOS was defined according to modified National Institutes of Health [NIH] 1990 criteria. ). Prediabetic hyperglycemia was determined by a 75-gram OGTT and included impaired fasting glucose (IFG), IGT, or both (IFG/IGT).
Pre-assignment Details: Exclusion criteria included diabetic subjects, smokers, suspected pregnancy, desiring pregnancy or injectable hormonal contraceptive use within 6 months; and use of oral contraceptives, other steroid hormones, drugs that affect gastrointestinal motility or carbohydrate metabolism and/or anti-obesity drugs within 3 months prior to study entry.
Groups:
- Metformin XR: Metformin 2000 mg QD for 16 weeks
  Metformin XR: Start 2 pills (2 pills of 500 mg =1000mg XR) for 3 weeks
  Increase to 4 pills as tolerated (4 pills of 500 mg XR =2000 mg XR) for remainder of study
- Saxagliptin: Saxagliptin 5 mg QD for 16 weeks
  Saxagliptin: Start 1 pill (5 mg)) for 3 weeks
  Remain at 1 pill (5mg dose) for remainder of study
- Saxagliptin-Metformin XR: Saxagliptin-Metformin XR (combination pill)
  5mg Saxagliptin/2000 mg Metformin XR QD for 16 weeks
  Saxagliptin-Metformin XR: Start 1 pill (2.5 mg/ 1000mg XR) for 3 weeks
  Increase to 2 pills as tolerated (5mg/2000 mg XR) for remainder of study
Period: Overall Study
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Started | 13 | 12 | 13
Completed | 12 | 11 | 11
Not Completed | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Noncompliant | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants had PCOS and were glucose impaired
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR | Total
Number analyzed (Participants) | 13 | 12 | 13 | 38
Age, Categorical [Count of Participants; unit: Participants] — All participants had to be 18 to 42 years to participate
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 13 | 12 | 13 | 38
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — All participants had to be female to qualify
  Participants
    Female | 13 | 12 | 13 | 38
    Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Our patient population is approximately 64% Caucasian and 35% African -American. The remaining ethnicities comprise about 1%.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 3 | 3 | 4 | 10
    White | 10 | 9 | 9 | 28
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — All participants were from Baton Rouge and surrounding parishes
  Participants
    United States | 13 | 12 | 13 | 38

OUTCOME MEASURES:

1. Primary Outcome: Glucose Metabolism
Description: Glucose metabolic secretory status after drug treatment (normal, impaired or diabetic). We used the American Diabetes Association (ADA) definition of impairment which is fasting glucose greater than 100 mg/dL and/or 2 hour glucose greater than 140 mg/dL.
Time Frame: 16 weeks
Population: Change from impaired to normal was evaluated. No patients were diabetic at the start or completion of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
Participants | 3 | 6 | 10
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin vs Saxagliptin-Metformin XR; Study change from dysglycemia to normal glucose state; Test type: Superiority or Other; p = .007, McNemar

2. Primary Outcome: Oral Disposition Index
Description: Post-treatment in insulin-sensitivity-secretion index . The insulin secretion-sensitivity index (IS-SI) provides an estimate of β-cell compensation relative to the prevailing insulin resistance, not absolute insulin secretion. It is derived by applying the concept of the disposition index (DI) to measurements obtained during the 2-h OGTT. The IS-SI, a surrogate measure of the DI derived from the OGTT (IGI multiplied by the SIOGTT], was calculated as the product of acute β-cell response [IGI] and Matsuda index (SIOGTT) based on the existence of the predicted hyperbolic relationship between these two measures
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
index | 208 (126) | 359 (295) | 532 (347)
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin vs Saxagliptin-Metformin XR; This was a Subjects (SS)/Groups repeated measures design; Test type: Superiority or Other; p = .02, ANOVA

3. Secondary Outcome: Fasting Glucose
Description: Post-treatment fasting glucose levels
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 5.4 (0.7) | 5.3 (.51) | 5.0 (.36)
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin vs Saxagliptin-Metformin XR; Pretreatment fasting glucose levels were compared with post-treatment levels; Test type: Superiority or Other; p < 0.0001, ANOVA; n

4. Secondary Outcome: Mean Blood Glucose During the OGTT
Description: Post-treatment mean blood glucose levels. Mean blood glucose (MBG) concentrations were calculated by summing glucose values obtained at 0,30,60 and 120 minutes during the OGTT and dividing by 4.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 7.9 (1.4) | 7.1 (1.64) | 6.2 (1.2)
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin vs Saxagliptin-Metformin XR; Test type: Superiority or Other; p = .038, ANOVA

5. Secondary Outcome: Matsuda Index of Insulin-Sensitivity (SI OGTT)
Description: Post-treatment insulin sensitivity index. The Matsuda index of whole-body insulin sensitivity is calculated from an oral glucose tolerance test (10,000/square root of [fasting glucose x fasting insulin] x [mean glucose x mean insulin during OGTT]), and is highly correlated with the rate of whole-body glucose disposal during the euglycemic insulin clamp
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
Index | 2.5 (1.6) | 3.5 (3.4) | 4.1 (2.6)
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin vs Saxagliptin-Metformin XR; Test type: Superiority or Other; p = 0.003, ANOVA

6. Secondary Outcome: Pancreatic ß-cell Compensatory Function
Description: Post-treatment corrected early phase insulin secretion index (IGI/HOMA-IR). . Early pancreatic β-cell response is estimated as the insulinogenic index (IGI) derived from the ratio of the increment of insulin to that of glucose 30 minutes after a glucose load (insulin 30 min - insulin 0 min/glucose 30 min - glucose 0 min) corrected for by the relative level of insulin resistance (IGI/HOMA-IR which is estimated by homeostasis model assessment of insulin resistance using fasting insulin and glucose levels).
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
Ratio | 0.46 (0.3) | 1.4 (1.7) | 1.03 (0.7)
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin vs Saxagliptin-Metformin XR; Test type: Superiority or Other; p = .025, ANOVA

7. Secondary Outcome: Body Mass Index at 16 Weeks
Description: Height and weight measurements were used to calculate body mass index (BMI), defined as kg/m2.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: kg/mg2
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
kg/mg2 | 42 (7.7) | 36.7 (7.4) | 42 (10.2)
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin vs Saxagliptin-Metformin XR; Test type: Superiority or Other; p = 0.006, ANOVA

8. Secondary Outcome: Waist Circumference at 16 Weeks
Description: The circumference measurement was taken in the upright position using a 15-mm width flexible metric tape held close to the body but not tight enough to indent the skin. Waist circumference (WC) was measured in centimeters at the narrowest level midway between the lowest ribs and the iliac crest.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
centimeters | 109 (13) | 99.6 (17) | 106 (16)
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin vs Saxagliptin-Metformin XR; Test type: Superiority or Other; p = .006, ANOVA

9. Secondary Outcome: Menstrual Cycle Interval at 16 Weeks
Description: The number of menstrual cycles during the previous year was recorded and the average menstrual interval calculated by dividing 365 by the number of menstrual cycles in the previous year . During the study period, the patients in a menstrual diary recorded vaginal bleeding over 16 weeks. The effects of treatment intervention on menstrual cycle interval was calculated evaluated by dividing 112 days by the number of menstrual cycles recorded in each patient's menstrual cycle diary.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: days between menstrual cycles
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
days between menstrual cycles | 81 (44) | 58 (29) | 36 (11)
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin vs Saxagliptin-Metformin XR; Test type: Superiority or Other; p = .026, ANOVA

10. Secondary Outcome: Triglyceride (TRG) /HDL-cholesterol Ratio
Description: The measure of TRG levels and HDL- cholesterol levels are used as an estimate of insulin sensitivity. A TRG/HDL-C ratio of greater than 3.0 is used as an indirect measure of insulin resistance
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
Ratio | 4.2 (2.4) | 2.9 (1.3) | 3.0 (0.9)
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin vs Saxagliptin-Metformin XR; Test type: Superiority or Other; p = .006, ANOVA

11. Secondary Outcome: Free Androgen Index (FAI)
Description: Hyperandrogenism is measured by a combination of total testosterone (T) and sex hormone binding globulin (SHBG). The FAI was calculated as the quotient 100 x T/SHBG; hyperandrogenism was defined by a FAI value >3.85.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
index | 6.3 (2.8) | 5.5 (3.4) | 4.3 (3.5)
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin; Test type: Superiority or Other; p = .006, ANOVA

12. Other Pre Specified Outcome: Number of Participants With No Clinically Significant Changes in Liver Enzyme Levels or Positive Pregnancy Tests
Description: The safety criteria will include laboratory values for liver enzymes and document the absence of pregnancy in all participants during the trial
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Number analyzed (Participants) | 12 | 11 | 11
Participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: Metformin XR vs Saxagliptin vs Saxagliptin-Metformin XR; Test type: Superiority or Other; p > 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: 22 months
Arm/Group | Metformin XR | Saxagliptin | Saxagliptin-Metformin XR
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 1/13 | 0/12 | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin XR (N=13) | Saxagliptin (N=12) | Saxagliptin-Metformin XR (N=13)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) — Common finding with metformin

LIMITATIONS AND CAVEATS:
Study limitations were the small number of patients and the short interval (16 weeks) of drug treatment.

Surrogate measures derived from the OGTT were used to estimate insulin sensitivity and secretion. .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes